CLINICAL TRIAL: NCT01171703
Title: Optimized Strategy for Diabetic Patients With Critical Limb Ischemia: A Multi-center, Randomized Controlled Trial and Registration Study(Part I)
Brief Title: Optimized Strategy for Diabetic Patients With Critical Limb Ischemia(Part I)
Acronym: DCLI-I
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liu Chang-wei, Vascular Surgery, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pumch-DCLI-I
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2010-07

CONDITIONS: Vascular Diseases; Diabetes
Keywords: Critical limb ischemia; Diabetes; Femoropopliteal artery bypass; Stent
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus; Chronic Limb-Threatening Ischemia | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bypass (Experimental): femoral-popliteal bypass
  Interventions: Device: femoral-popliteal bypass
- stent (Experimental)
  Interventions: Device: stent

INTERVENTIONS:
Device: femoral-popliteal bypass — Before operation, take aspirin 100mg every day. Groin and suprageniculate incision, PTFE graft with end to side anastomoses.
  Arms: bypass
Device: stent — Before operation, take aspirin 100mg every day. During the operation, stent is delivered by a catheter and positioned through the narrowing in the artery. The stent is then expanded against the wall of the blood vessel to provide a wider channel for blood. At last, use balloon dilate the stent.
  Arms: stent

SUMMARY:
The purpose of this trial is to find out the appropriate way to treat DM patients with critical limb ischemia. This trial includes two parts. Part I focuses on the treatment of femoral arterial lesion and part II focuses on the treatment of below-knee arterial lesion.

DETAILED DESCRIPTION:
The trial includes two parts and here is part I. This part is a multi-center, prospective, randomized, controlled study to compare the therapeutic effect of stent and bypass to chronic long occlusion of the superficial femoral artery in DM patients. Totally 70 patients will be entered into the study. The lesion of the femoral artery should be TASC B、C or D and the patients should suffered ischemic symptom with Rutherford 3-6.The lesion does not extend beyond the aortoiliac artery or blow-knee popliteal artery, with at least 1 vessel infra-popliteal runoff to the foot.

ELIGIBILITY:
Inclusion Criteria:

* The patients volunteer to join the trial and sign the formal consent.
* The patients are ≥55 year-old and ≤75 year-old.
* The patients suffer from symptomatic leg ischemia with rutherford classification3, 4 , 5 or 6. The presentation is severe intermittent claudication, rest pain, ulcer or gangrene.
* The lesion of the femoral artery should be TASC B、C or D.
* The femoral-popliteal artery has never received bypass or endovascular therapy before.
* No obvious stenosis or occlusion in the aortoiliac artery; or the lesion could be treated simultaneously or has already been cured.
* No obvious stenosis in below-knee popliteal artery; at least 1 vessel infra-popliteal runoff to the foot.
* No surgical contraindications;no infection in operation region.
* Be diagnosed with DM for at least 1 year.

Exclusion Criteria:

* Refuse random treatment.
* Previous operations on the superficial femoral artery.
* Acute lower extremity arterial thrombosis.
* Serious major organ failure.
* Allergic to the contrast agent or has contrast nephropathy.
* No clinical compliance or unfit to join the trial

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Occlusion of the stent or bypass | 36 months

SECONDARY OUTCOMES:
Mortality | 30 days
  The number of death during the first month after procedure, no matter whether the cause of death is related to the procedure.
Rate of limb salvage | 36 months
Procedural complications, defined as any adverse event | 36 months
  including MI, DVT, hematoma, renal failure, wound infection, lymphatic fistula
Quality of Life assessment | 36 months
  assessment in 1 month,6 months,12 months,24 months and 36 months post procedure
Restenosis measured by Duplex Ultrasound or CTA | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Liu changwei, bachelor, Study Chair
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Beijing, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality

REFERENCES:
- See also: the website of the vascular surgery department of PUMCH — http://www.vascular.cn/